CLINICAL TRIAL: NCT02000076
Title: The Stockholm Sleepy Brain Study: Effects of Sleep Deprivation on Cognitive and Emotional Processing in Young and Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mats Lekander (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor-Investigator, Mats Lekander, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Sleepy Brain Study Wave 1
Record Dates: First submitted 2013-08-13; First posted 2013-12-03 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Deprivation
Keywords: Sleep; resting state; functional connectivity; emotional contagion; empathy; emotional regulation
MeSH Terms: conditions — Sleep Deprivation; Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep deprivation (Experimental): Partial sleep deprivation allowing 3 h sleep at night
  Interventions: Behavioral: Partial sleep deprivation allowing 3 h sleep at night
- Full sleep (Experimental): Sleep with no restriction
  Interventions: Behavioral: Full sleep

INTERVENTIONS:
Behavioral: Partial sleep deprivation allowing 3 h sleep at night — Participants sleep at home while monitored with ambulatory polysomnography. For the full sleep condition, they are instructed to go to bed and to get up at the usual times that they would normally do that. For the sleep deprivation condition, they are instructed to go to bed 3 hours before the time when they would usually get up, and then to get up at that time.
  Other Names: Sleep restriction; Sleep loss
  Arms: Sleep deprivation
Behavioral: Full sleep — Participants sleep at home while monitored with ambulatory polysomnography. For the full sleep condition, they are instructed to go to bed and to get up at the usual times that they would normally do that. For the sleep deprivation condition, they are instructed to go to bed 3 hours before the time when they would usually get up, and then to get up at that time.
  Arms: Full sleep

SUMMARY:
The main purpose of this study is to investigate the effects of partial sleep deprivation (PSD) on resting state brain connectivity, emotional contagion, empathy, and emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years of age, inclusive OR 65-75 years of age, inclusive
* Able to understand spoken and written Swedish (in order to understand instructions)
* Normal or corrected-to-normal vision not using glasses
* Not colour blind
* Right-handed
* Free from ferromagnetic objects in body
* No history of any neurologic or psychiatric illness including drug abuse
* No history of diabetes nor hypertension

  * No depression according to ratings using the Hospital Anxiety and Depression scale (HAD)
  * No insomnia according to ratings using the Insomnia Severity Index (ISI) and Karolinska Sleep Questionnaire (KSQ)
* No use of psychotropic drugs
* Not studying or working in medicine, psychology, nor behavioural science
* Not suffering from severe seasonal allergy
* No use of cortisone, anti-histamines, nor any other immune-modulating drugs
* Habitual intake of no more than 4 cups of coffee per day or the equivalent in terms of caffeine
* No daily use of nicotine

Exclusion Criteria:

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level-dependent response in amygdala to angry faces (t/z-score from statistical parametric mapping) | Change between 1st and 2nd MRI scanning session (approx. 1 month later)
  This registration is made in order to pre-specify hypotheses in a basic science project. For a full list of outcomes and hypotheses, see study description (above).

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Åkerstedt, PhD, Study Chair — Stockholm University; Mats Lekander, PhD, Principal Investigator — Stockholm University, Karolinska Institutet; Håkan Fischer, PhD, Principal Investigator — Stockholm University
Locations (1):
- Karolinska Institutet, Karolinska Universitetssjukhuset i Solna, Stockholm, None/Not Applicable, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared through the openfmri.org data repository.

REFERENCES:
- [Derived] Tamm S, Schwarz J, Thune H, Kecklund G, Petrovic P, Akerstedt T, Fischer H, Lekander M, Nilsonne G. A combined fMRI and EMG study of emotional contagion following partial sleep deprivation in young and older humans. Sci Rep. 2020 Oct 21;10(1):17944. doi: 10.1038/s41598-020-74489-9. PMID 33087746
- See also: List of hypotheses — https://osf.io/bxfsb/